CLINICAL TRIAL: NCT02998918
Title: Effects of Short-term Curcumin and Multi-polyphenol Supplementation on the Anti-inflammatory Properties of HDL
Acronym: PSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Mark Sarzynski, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00055882
Record Dates: First submitted 2016-10-18; First posted 2016-12-21 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Inflammation; Atherosclerosis; Cardiovascular Disease
Keywords: Inflammation; HDL; Anti-inflammatory; Supplementation; Curcumin; polyphenol; V-cam; I-cam; atherosclerosis; cardiovascular disease; atherogenesis; antioxidant; resveratrol; quercetin
MeSH Terms: conditions — Inflammation; Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PolyResveratrol Supplementation (Experimental): Participants take 500 mg of PolyResveratrol (100 mg curcumin phytosome, 100 mg quercetin phytosome, 100 mg green tea phytosome, 100 mg trans-resveratrol, 100 mg trans-pterostilbene; Thorne Research) twice daily for one week. Two blood Draws are taken on both the first and last days of the week. One blood draw is done fasted just before consumption of one supplement dose, and one blood draw is done after consumption of one supplement dose.
  Interventions: Dietary Supplement: PolyResveratrol Supplementation
- Curcumin Supplementation (Experimental): Participants take 500 mg of Curcumin phytosome twice daily for one week. Two blood draws are taken on both the first and last days of the week. One blood draw is done fasted just before consumption of one supplement dose, and one blood draw is done after consumption of one supplement dose.
  Interventions: Dietary Supplement: Curcumin Supplementation

INTERVENTIONS:
Dietary Supplement: PolyResveratrol Supplementation — Participants will take 1 mg of a polyresveratrol phytosome supplement each day for one week. The acute effect (1 hr) of one 500 mg dose of the polyresveratrol phytosome supplement on inflammation will be examined along with the short-term effect (1 week).
  Arms: PolyResveratrol Supplementation
Dietary Supplement: Curcumin Supplementation — Participants will take 1 mg of a curcumin phytosome supplement each day for one week. The acute effect (1 hr) of one 500 mg dose of the curcumin phytosome supplement on inflammation will be examined along with the short-term effect (1 week).
  Arms: Curcumin Supplementation

SUMMARY:
Polyphenol supplements, including curcumin and resveratrol, are known to decrease inflammation, but previous polyphenol supplements were poorly absorbed and thus their effects were reduced. A new phytosome formulation coats the supplements and allows them to be better absorbed. The purpose of this study is to examine the acute (1-hr) and short-term (1-week) effects of two different phytosome-formulated polyphenol supplements on inflammation. The two supplements that will be used are: 1) PolyResveratrol and 2) Curcumin.

DETAILED DESCRIPTION:
Atherosclerosis is a chronic inflammatory disease underlying coronary artery disease, driven in part by the innate immune system, particularly macrophages. The adhesion of leukocytes to the vascular endothelium, mediated by endothelial cellular adhesion molecules including vascular adhesion molecule-1 (VCAM-1) and intercellular adhesion molecule-1 (ICAM-1), is one of the crucial initial steps in atherogenesis. Elevated levels of high-density lipoprotein cholesterol (HDL-C) are associated with reduced risk for cardiovascular disease (CVD); however, interventions designed to increase HDL-C concentration in humans have yet to lead to reductions in cardiovascular events. A possible explanation for the failure of recent clinical trials is the structural and functional complexity of HDL particles, which have multiple cardioprotective properties, including anti-inflammatory, antioxidative, and reverse cholesterol transport activities. The anti-inflammatory effects of HDL include reduction of inflammatory cytokines and vascular leukocyte adhesion molecules. A recent study showed that dietary composition can affect HDL's anti-inflammatory properties, namely the ability to inhibit the expression of ICAM-1 and VCAM-1.

Numerous studies have shown that polyphenols, including curcumin, quercetin, and resveratrol, exhibit multiple health benefits, including anti-inflammatory properties. Curcumin is a flavonoid polyphenol that is the active ingredient in the spice turmeric. Quercetin is one of the most abundant dietary flavonoids and is found in many fruits, vegetables, and beverages. Resveratrol is a non-flavonoid polyphenol present in a limited number of plant-derived foods, including grapes and peanuts. In vitro studies show these three polyphenols independently decrease VCAM-1 and ICAM-1 expression induced by tumor necrosis factor alpha (TNFα) in human endothelial cells, as well as increase cholesterol efflux to apolipoprotein A-I (apoA-I) and HDL in macrophages. However, previous in vitro models used direct incubation with each polyphenol (i.e., HDL was directly exposed to the polyphenol in the cell culture, as opposed to incubation with plasma after consumption of the polyphenol), with doses much higher than found in typical human diets or supplements.

The health effects of polyphenols in humans are limited by their poor bioavailability, as they are rapidly metabolized and excreted. Recent studies have found that formulating poorly-absorbed molecules with phosphatidylcholine via phytosomes increases their bioavailability. For example, recent studies comparing curcumin phytosome (Meriva®) and standard curcumin formulations in humans found that the curcumin phytosome formulation increased curcuminoid bioavailability between 8- to 29-fold. To our knowledge, no study has examined the effects of polyphenol supplementation, particularly phytosome-formulated polyphenols, in humans on the ability of circulating plasma to inhibit the expression of cellular adhesion molecules or enhance cholesterol efflux capacity in vitro. Furthermore, it is unknown whether polyphenol supplementation modulates the ability of HDL particles to perform these same functions.

Therefore, the purpose of this study is to examine whether acute and short-term (1-week) polyphenol supplementation in humans affects inflammation measured at the whole plasma level, as well as the inflammatory and cholesterol efflux properties of HDL particles. The investigators will test the effects of two supplements in a cross-over design: a curcumin phytosome and a multi-polyphenol supplement (containing curcumin phytosome, quercetin phytosome, and trans-resveratrol). The investigators hypothesize that one of the mechanisms by which polyphenols exert a beneficial effect on inflammation and atherosclerosis is through its modulation of HDL particles.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* Between 18 and 60 years old
* Non-smoker
* Not taking any medications or dietary supplements

Exclusion Criteria:

* Taking prescription anti-inflammatory drugs or supplements/drugs that may affect inflammation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sarzynski, Principal Investigator — University of South Carolina
Locations (1):
- Clinical Exercise Research Center, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Seneviratne AN, Sivagurunathan B, Monaco C. Toll-like receptors and macrophage activation in atherosclerosis. Clin Chim Acta. 2012 Jan 18;413(1-2):3-14. doi: 10.1016/j.cca.2011.08.021. Epub 2011 Aug 22. PMID 21884686
- [Background] Emerging Risk Factors Collaboration; Di Angelantonio E, Sarwar N, Perry P, Kaptoge S, Ray KK, Thompson A, Wood AM, Lewington S, Sattar N, Packard CJ, Collins R, Thompson SG, Danesh J. Major lipids, apolipoproteins, and risk of vascular disease. JAMA. 2009 Nov 11;302(18):1993-2000. doi: 10.1001/jama.2009.1619. PMID 19903920
- [Background] Toth PP, Barter PJ, Rosenson RS, Boden WE, Chapman MJ, Cuchel M, D'Agostino RB Sr, Davidson MH, Davidson WS, Heinecke JW, Karas RH, Kontush A, Krauss RM, Miller M, Rader DJ. High-density lipoproteins: a consensus statement from the National Lipid Association. J Clin Lipidol. 2013 Sep-Oct;7(5):484-525. doi: 10.1016/j.jacl.2013.08.001. Epub 2013 Aug 11. PMID 24079290
- [Background] Barter PJ, Nicholls S, Rye KA, Anantharamaiah GM, Navab M, Fogelman AM. Antiinflammatory properties of HDL. Circ Res. 2004 Oct 15;95(8):764-72. doi: 10.1161/01.RES.0000146094.59640.13. PMID 15486323
- [Background] Nicholls SJ, Lundman P, Harmer JA, Cutri B, Griffiths KA, Rye KA, Barter PJ, Celermajer DS. Consumption of saturated fat impairs the anti-inflammatory properties of high-density lipoproteins and endothelial function. J Am Coll Cardiol. 2006 Aug 15;48(4):715-20. doi: 10.1016/j.jacc.2006.04.080. Epub 2006 Jul 24. PMID 16904539
- [Background] Bisht K, Wagner KH, Bulmer AC. Curcumin, resveratrol and flavonoids as anti-inflammatory, cyto- and DNA-protective dietary compounds. Toxicology. 2010 Nov 28;278(1):88-100. doi: 10.1016/j.tox.2009.11.008. Epub 2009 Nov 10. PMID 19903510
- [Background] Hatcher H, Planalp R, Cho J, Torti FM, Torti SV. Curcumin: from ancient medicine to current clinical trials. Cell Mol Life Sci. 2008 Jun;65(11):1631-52. doi: 10.1007/s00018-008-7452-4. PMID 18324353
- [Background] Strimpakos AS, Sharma RA. Curcumin: preventive and therapeutic properties in laboratory studies and clinical trials. Antioxid Redox Signal. 2008 Mar;10(3):511-45. doi: 10.1089/ars.2007.1769. PMID 18370854
- [Background] Smoliga JM, Baur JA, Hausenblas HA. Resveratrol and health--a comprehensive review of human clinical trials. Mol Nutr Food Res. 2011 Aug;55(8):1129-41. doi: 10.1002/mnfr.201100143. Epub 2011 Jun 20. PMID 21688389
- [Background] Tome-Carneiro J, Larrosa M, Gonzalez-Sarrias A, Tomas-Barberan FA, Garcia-Conesa MT, Espin JC. Resveratrol and clinical trials: the crossroad from in vitro studies to human evidence. Curr Pharm Des. 2013;19(34):6064-93. doi: 10.2174/13816128113199990407. PMID 23448440
- [Background] Boots AW, Haenen GR, Bast A. Health effects of quercetin: from antioxidant to nutraceutical. Eur J Pharmacol. 2008 May 13;585(2-3):325-37. doi: 10.1016/j.ejphar.2008.03.008. Epub 2008 Mar 18. PMID 18417116
- [Background] Russo M, Spagnuolo C, Tedesco I, Bilotto S, Russo GL. The flavonoid quercetin in disease prevention and therapy: facts and fancies. Biochem Pharmacol. 2012 Jan 1;83(1):6-15. doi: 10.1016/j.bcp.2011.08.010. Epub 2011 Aug 16. PMID 21856292
- [Background] Ferrero ME, Bertelli AE, Fulgenzi A, Pellegatta F, Corsi MM, Bonfrate M, Ferrara F, De Caterina R, Giovannini L, Bertelli A. Activity in vitro of resveratrol on granulocyte and monocyte adhesion to endothelium. Am J Clin Nutr. 1998 Dec;68(6):1208-14. doi: 10.1093/ajcn/68.6.1208. PMID 9846848
- [Background] Binion DG, Heidemann J, Li MS, Nelson VM, Otterson MF, Rafiee P. Vascular cell adhesion molecule-1 expression in human intestinal microvascular endothelial cells is regulated by PI 3-kinase/Akt/MAPK/NF-kappaB: inhibitory role of curcumin. Am J Physiol Gastrointest Liver Physiol. 2009 Aug;297(2):G259-68. doi: 10.1152/ajpgi.00087.2009. Epub 2009 Jun 11. PMID 19520742
- [Background] Kleemann R, Verschuren L, Morrison M, Zadelaar S, van Erk MJ, Wielinga PY, Kooistra T. Anti-inflammatory, anti-proliferative and anti-atherosclerotic effects of quercetin in human in vitro and in vivo models. Atherosclerosis. 2011 Sep;218(1):44-52. doi: 10.1016/j.atherosclerosis.2011.04.023. Epub 2011 May 5. PMID 21601209
- [Background] Berrougui H, Grenier G, Loued S, Drouin G, Khalil A. A new insight into resveratrol as an atheroprotective compound: inhibition of lipid peroxidation and enhancement of cholesterol efflux. Atherosclerosis. 2009 Dec;207(2):420-7. doi: 10.1016/j.atherosclerosis.2009.05.017. Epub 2009 May 22. PMID 19552907
- [Background] Voloshyna I, Hai O, Littlefield MJ, Carsons S, Reiss AB. Resveratrol mediates anti-atherogenic effects on cholesterol flux in human macrophages and endothelium via PPARgamma and adenosine. Eur J Pharmacol. 2013 Jan 5;698(1-3):299-309. doi: 10.1016/j.ejphar.2012.08.024. Epub 2012 Oct 4. PMID 23041272
- [Background] Chen FY, Zhou J, Guo N, Ma WG, Huang X, Wang H, Yuan ZY. Curcumin retunes cholesterol transport homeostasis and inflammation response in M1 macrophage to prevent atherosclerosis. Biochem Biophys Res Commun. 2015 Nov 27;467(4):872-8. doi: 10.1016/j.bbrc.2015.10.051. Epub 2015 Oct 19. PMID 26471308
- [Background] Chang YC, Lee TS, Chiang AN. Quercetin enhances ABCA1 expression and cholesterol efflux through a p38-dependent pathway in macrophages. J Lipid Res. 2012 Sep;53(9):1840-50. doi: 10.1194/jlr.M024471. Epub 2012 Jun 18. PMID 22711909
- [Background] Cuomo J, Appendino G, Dern AS, Schneider E, McKinnon TP, Brown MJ, Togni S, Dixon BM. Comparative absorption of a standardized curcuminoid mixture and its lecithin formulation. J Nat Prod. 2011 Apr 25;74(4):664-9. doi: 10.1021/np1007262. Epub 2011 Mar 17. PMID 21413691
- [Background] Jager R, Lowery RP, Calvanese AV, Joy JM, Purpura M, Wilson JM. Comparative absorption of curcumin formulations. Nutr J. 2014 Jan 24;13:11. doi: 10.1186/1475-2891-13-11. PMID 24461029
- [Background] Gordon SM, Deng J, Lu LJ, Davidson WS. Proteomic characterization of human plasma high density lipoprotein fractionated by gel filtration chromatography. J Proteome Res. 2010 Oct 1;9(10):5239-49. doi: 10.1021/pr100520x. PMID 20718489
- [Background] Cockerill GW, Rye KA, Gamble JR, Vadas MA, Barter PJ. High-density lipoproteins inhibit cytokine-induced expression of endothelial cell adhesion molecules. Arterioscler Thromb Vasc Biol. 1995 Nov;15(11):1987-94. doi: 10.1161/01.atv.15.11.1987. PMID 7583580

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: PolyResveratrol Then Curcumin Supplementation: Week 1 Polyresveratrol supplementation: Group 1 participants take 500 mg of PolyResveratrol (100 mg curcumin phytosome, 100 mg quercetin phytosome, 100 mg green tea phytosome, 100 mg trans-resveratrol, 100 mg trans-pterostilbene; Thorne Research) twice daily for one week. The acute effect (1 hr) of one 500 mg dose of the polyresveratrol phytosome supplement on inflammation will be examined along with the short-term effect (1 week).
  Weeks 2-3 Washout period: After the one week polyresveratrol supplementation period, the subjects go through a 2-week washout period with no supplementation.
  Week 4 Curcumin supplementation: In this cross-over trial, group 1 participants take 500 mg of Curcumin phytosome twice daily for one week during week 4. The acute effect (1 hr) of one 500 mg dose of the curcumin phytosome supplement on inflammation will be examined along with the short-term effect (1 week).
- Group 2: Curcumin Followed by Polyresveratrol Supplementation: Week 4 Curcumin supplementation: Group 2 participants take 500 mg of Curcumin phytosome twice daily for one week. The acute effect (1 hr) of one 500 mg dose of the curcumin phytosome supplement on inflammation will be examined along with the short-term effect (1 week).
  Weeks 2-3 Washout period: After the one week Curcumin supplementation period, the subjects go through a 2-week washout period with no supplementation.
  Week 4 Polyresveratrol supplementation: Group 2 participants take 500 mg of PolyResveratrol (100 mg curcumin phytosome, 100 mg quercetin phytosome, 100 mg green tea phytosome, 100 mg trans-resveratrol, 100 mg trans-pterostilbene; Thorne Research) twice daily for one week during the 4th week of the study. The acute effect (1 hr) of one 500 mg dose of the polyresveratrol phytosome supplement on inflammation will be examined along with the short-term effect (1 week).
Period: Overall Study
Arm/Group | Group 1: PolyResveratrol Then Curcumin Supplementation | Group 2: Curcumin Followed by Polyresveratrol Supplementation
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: PolyResveratrol Then Curcumin Supplementation: Group 1 consumed 1 mg/day (one dose of 500 mg/two capsules in morning and two capsules/500 mg at night) of Polyresveratrol-SR for one week in phase 1 then after a 2-week washout period consumed 1 mg/day (one dose of 500 mg/two capsules in morning and one dose of 500 mg at night) of Meriva 500-SF (curcumin phytosome) for one week during phase 2 of the crossover trial
- Group 2: Curcumin Then PolyResveratrol Supplementation: Group 2 consumed 1 mg/day (one dose of 500 mg/two capsules in morning and two capsules/500 mg at night) of Meriva 500-SF (curcumin phytosome) for one week in phase 1 then after a 2-week washout period consumed 1 mg/day (one dose of 500 mg/two capsules in morning and one dose of 500 mg at night) of Polyresveratrol-SR for one week during phase 2 of the crossover trial
- Total: Total of all reporting groups
Arm/Group | Group 1: PolyResveratrol Then Curcumin Supplementation | Group 2: Curcumin Then PolyResveratrol Supplementation | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (6.3) | 30.0 (7.4) | 28.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.2 (4.5) | 25.0 (5.0) | 24.4 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Inflammation Change: HDL Plasma
Description: VCAM-1 expression in HDL plasma will be measured at baseline, and after one week of supplementation for each supplement. Differences in one-week changes in inflammation between each supplement will be compared.
Time Frame: One week
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | Group 1: PolyResveratrol Then Curcumin Supplementation | Group 2: Curcumin Then PolyResveratrol Supplementation
Number analyzed (Participants) | 11 | 10
AU | NA (NA) — The assays for this measure would not produce valid/reliable results on our stored specimens. Thus, we will not be reporting data for this outcome. | NA (NA) — The assays for this measure would not produce valid/reliable results on our stored specimens. Thus, we will not be reporting data for this outcome.

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the start of the study until 4 weeks later.
Groups:
- PolyResveratrol Supplementation: 1 mg/day (one dose of 500 mg/two capsules in morning and two capsules/500 mg at night) of Polyresveratrol-SR for one week
- Curcumin Supplementation: 1 mg/day (one dose of 500 mg/two capsules in morning and two capsules/500 mg at night) of Meriva 500-SF (curcumin phytosome) for one week
Arm/Group | PolyResveratrol Supplementation | Curcumin Supplementation
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
The planned assays did not work in the stored specimens. Thus, data will not be reported for this trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT02998918/Prot_SAP_000.pdf